CLINICAL TRIAL: NCT06021522
Title: A Multicenter, Open-Label, Study to Evaluate the Long-term Safety of Ecopipam Tablets in Children, Adolescents and Adults With Tourette's Disorder
Brief Title: A Study to Evaluate Long-term Safety of Ecopipam Tablets in Children, Adolescents and Adults With Tourette's Disorder
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBS-101-TD-391; 2023-503545-67-00 (Other: EUCT)
Record Dates: First submitted 2023-07-11; First posted 2023-09-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Tourette Syndrome
Keywords: Ecopipam; Neurodevelopmental Disorders; Mental Disorders; Central Nervous System Depressants; Neurodegenerative Diseases; Movement Disorders; Tic Disorders; Nervous System Diseases; Central Nervous System Diseases; Brain Diseases
MeSH Terms: conditions — Tourette Syndrome; Neurodevelopmental Disorders; Mental Disorders; Neurodegenerative Diseases; Movement Disorders; Tic Disorders; Nervous System Diseases; Central Nervous System Diseases; Brain Diseases | interventions — ecopipam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ecopipam 1.8 mg/kg/day (Experimental): Ecopipam tablets will be administered orally (PO) once daily in the evening without regard to meals at concentrations 11.2, 22.4, 33.6, 44.8, 67.2 and 89.6 milligrams (mg) containing 12.5, 25, 37.5, 50, 75 and 100 mg ecopipam HCl, respectively in 4-week titration phase to achieve a target dose of 1.8 milligram per kilogram per day (mg/kg/day) ecopipam (2 mg/kg/day ecopipam HCl). Participants will be evaluated for safety at each baseline visit and at all treatment visits up to 24 months and at follow up visits at 7 and 14 days after last dose of ecopipam.
  Interventions: Drug: Ecopipam

INTERVENTIONS:
Drug: Ecopipam — Selective dopamine D1 and D5 receptor antagonist
  Other Names: Ecopipam Hydrochloride

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of ecopipam tablets in children (greater than or equal to [>=] 6 and less than [<] 12 years of age), adolescents (>=12 and <18 years of age), and adults (>=18 years of age) with Tourette's Syndrome (TS).

DETAILED DESCRIPTION:
This study is to evaluate the long-term safety and tolerability of ecopipam tablets in eligible participants. The eligible participants will be entered into a treatment period and start a 4-week titration phase to achieve a target steady-state dose of 1.8 milligram per kilogram per day (mg/kg/day) ecopipam (2 mg/kg/day dose of ecopipam HCl). During the 4-week titration phase ecopipam will be dispensed following weight bands before reaching their respective maintenance dose until end of the treatment. Safety assessment will be conducted at baseline visit and at all treatment visits (Months 1-12, 15, 18, 21 and 24). Safety follow up visits will be conducted 7 and 14 days and a follow up phone call will be conducted 30 days after the last dose of ecopipam.

ELIGIBILITY:
Inclusion Criteria:

* >=6 to >=18 years of age.
* Participants enrolling from the study EBS-101-TD-301; completed all visits through Week 24 and days 7 and 14 safety follow-up, met relapse criteria during the double-blind randomized (R/WD) period after completing the 301 end of trial (ET) visit, the 7 day and 14 day safety follow up visits, but not before 24 weeks following the 301 baseline visit or participants who met relapse criteria will be eligible after completing early termination visit, Day 7 and Day 14 follow up visits.
* Participants who completed the studies EBS-101-OL-001 or PSY302A.
* The enrolling participant must have had clinical benefit from ecopipam and would benefit from continued participation.
* Effective contraception during the study and 30 days after last study dose for sexually active participants
* <18 years of age participants parent/legal guardian must sign a written informed consent and participant must sign a written informed assent.
* Participant must have TD based on Diagnostic and Statistical Manual for Mental Disorders - 5th Edition (DSM-5-TR diagnostic criteria) for TD.
* TD diagnosis and both motor and vocal tics that cause impairment with normal routines

Exclusion Criteria:

* The participants who discontinued the studies PSY-302A, EBS-101-OL-001 or EBS-101-TD-301 due to reasons such as either lost to follow up, withdrawn consent, non-compliant or withdrawn by the discretion of either the site investigator or the sponsor.
* Participants with ongoing or past history of neurological condition (example [e.g.], Huntington's disease, Parkinson's disease, Wilson's disease, stroke, Restless Legs Syndrome).
* Any unstable mood disorder (DSM-5-TR criteria), mental illness or clinically significant lab abnormalities, moderate to severe renal or hepatic impairment, a PHQ-9 score >=10 at screening and history of neuroleptic malignant syndrome at the time of screening or baseline.
* Participants who completed the studies EBS-101-OL-001 or PSY-302A and who had previous exposure to ecopipam and oral neuroleptics within 4 weeks and depot neuroleptics within 3 months prior to screening, 6 months prior to Baseline.
* Participants receiving any other medication to treat motor or vocal tics and anti-depressant or anti-anxiety medications.
* Risk of suicide as per PI judgement
* Pregnant or lactating women
* Certain medications that would have unfavorable drug interactions with ecopipam, e.g., digoxin, fluoxetine, valproic acid, bupropion.
* Current or recent (past 3 months) DSM-5-TR substance use disorder (with the exception of nicotine).
* Recent behavioral therapy
* Positive urine drug screen for cocaine, amphetamine, benzodiazepines, barbiturates, phencyclidine (PCP) or opiates at Baseline, except those receiving stable, prescribed treatment for attention deficit/hyperactivity disorder (ADHD)
* Lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any other psychotic disorder.
* Unable to swallow tablets.
* Known hypersensitivity to any of ecopipam's excipients.
* History of seizures (excluding febrile seizures that occurred >2 years prior to Baseline).
* Myocardial infarction within 6 months from Screening.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Baseline up to Month 24
  An adverse event (AE) is defined as any untoward medical occurrence in a subject administered a study drug and which does not necessarily have a causal relationship with this treatment. A TEAE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered casually related to the product.

CONTACTS AND LOCATIONS:
Locations (66):
- United States (43):
  - Harmonex, Inc., Dothan, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - CenExel CIT-IE, Bellflower, California
  - Cortica Site Network, Glendale, California
  - Cortica Site Network - San Rafael, San Rafael, California
  - Yale School of Medicine, New Haven, Connecticut
  - Childrens National Hospital, Washington D.C., District of Columbia
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Research in Miami Inc, Hialeah, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG Research, LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Lurie Children Hospital of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Josephson-Wallack-Munshower Neurology, Indianapolis, Indiana
  - University of Louisville Research Foundation Inc., Louisville, Kentucky
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts
  - Umass Chan Medical School, Worcester, Massachusetts
  - Michigan Clinical research Institute PC, Ann Arbor, Michigan
  - Neurobahavioral Medicine Group, Bloomfield Hills, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Alivation Research, Lincoln, Nebraska
  - University of Rochester, Rochester, New York
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - National Childrens Hospital - The Ohio State University, Columbus, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Providence Brain and Spine Institute, Portland, Oregon
  - Coastal Pediatric Research, Charleston, South Carolina
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Road Runner Research, Ltd, San Antonio, Texas
  - Cedar Clinical Research, Draper, Utah
  - Core Clinical Research, Everett, Washington
- Bulgaria (3):
  - Center Spectar-Plovdiv, Plovdiv, Bulgaria
  - ASMP-IP- d-r Kayryakova, Sofia, Sofia-Grad
  - Kalimat Medical Center_Sofia, Sofia
- The Kids Clinic Inc, Ajax, Ontario, Canada
- Hungary (2):
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Gyermek-es Ifjusagpszicihatria, Szeged, Hungary
  - Bethesda Childrens Hospital(Magyarországi Református Egyház Bethesda Gyermekkórháza), Budapest
- Italy (5):
  - Istituto Giannina Gaslini, Universita di Genova, Genova, GE
  - Universita degli Studi di Napoli Federico II, Napoli, Napoli
  - Ospedale Pediatrico Bambino Ges, Roma, RM
  - Azienda Ospedaliero Universitaria " G. Rodolico - San Marco", Catania
  - IRCCS Istituto Neurologico Carlo Besta, Milan
- Poland (5):
  - Neurologia Śląska Centrum Medyczne, Katowice, Poland
  - Gdanskie Centrum Zdrowia Sp z o.o., Gdansk, Pomeranian Voivodeship
  - Clinical Research Center Sp. z o.o. MEDIC-R Sp.k., Poznan, Wielkopolska
  - Wojewdzki Specjalistyczny Szpital Dziecicy im. sw. Ludwika w Krakowie, Krakow, Woj. Malopolskie
  - Centrum Medyczne Plejady, Krakow
- Serbia (3):
  - Institute of Mental Health, Belgrade, Belgrad
  - Clinic of Neurology and Psychiatry for Children and Adolescents, Belgrade, Grad Beograd
  - Clinical Centre Nis Center of Mental Health, Niš, Serbia
- Spain (4):
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No